CLINICAL TRIAL: NCT01267565
Title: Tracheal Dosage of Amylase : a New Surrogate for Microaspirations in Ventilated ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Victor Segalen Bordeaux 2 (Other)
Responsible Party: Principal Investigator, Alexandre Boyer, M.D., Université Victor Segalen Bordeaux 2
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ABoyer4
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Ventilated-acquired Pneumonia
Keywords: ventilator-acquired pneumonia; prevention; amylase; tracheal aspiration; microaspiration
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intubated and ventilated patients (Other): patients undergoing mechanical ventilation for an anticipated length of more than 48h
  Interventions: Other: dosage of amylase
- non intubated patients (Other): non intubated patients with an independant indication of bronchoscopy including an endotracheal aspiration during the procedure
  Interventions: Other: dosage of amylase

INTERVENTIONS:
Other: dosage of amylase — 4 sets of aspirations on one day per inclusion in the intubated and ventilated patients group and 1 set of aspiration in the non intubated patients group

SUMMARY:
Microaspirations of the oropharyngeal ± gastric contents through the endotracheal tube cuff contribute to the constitution of VAP. The pepsin has been recently proved effective as a surrogate of gastric content and was assessed in tracheal secretions. However, the pepsin dosage is fastidious, expensive and only characterizes aspirations from gastric origin. The aim of our study is to asses whether the value of amylase, which is mostly secreted by salivary glands, may turn out to be a new and simpler surrogate for microaspirations in ventilated ICU patients. Thirty patients ventilated for an anticipated length > 48h whose endotracheal tube includes a subglottic secretion device and producing sufficient endotracheal aspirations will be included. From H48, 4 sets of 3 aspirations each (oral, subglottic, tracheal) will be performed during one ventilation day for amylase dosage purpose. In ten of these patients, a comparison between pepsin and amylase will be assessed. In addition, 10 non intubated patients with an indication to bronchoscopy and necessitating a tracheal aspiration during the procedure will be included as a control group. The primary assessment criteria will be the oral/tracheal amylase ratio.

ELIGIBILITY:
Inclusion Criteria:

* intubated and ventlated patients group: patients ventilated with a tube including a subglottic secretion device for an anticipated length > 48h and producing sufficient endotracheal aspirations
* non intubated patients group: patients with an study-independant indication to bronchoscopy and necessitating a tracheal aspiration during the procedure

Exclusion Criteria:

* patients ventilated for less than 48h
* patients developing ventilated-acquired pneumonia or bronchitis before potential inclusion
* paralysed patients
* patients requiring a closed suction device
* patients with relative contraindications to endotracheal aspiration (status asthmaticus, severe ARDS with PF ratio < 100, hemorragic risk, brochopleural fistula)
* bronchiectasis, cystic fibrosis
* moribund patient or ethical decision to withhold or withdraw intensive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
oral/tracheal amylase ratio | up to 24h after bronchoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France